CLINICAL TRIAL: NCT05024630
Title: Renal Denervation and pUlmonary Vein isolAtion With cryoabLation on Atrial fIbrillation reCurrence Among Patients With Paroxysmal Atrial Fibrillation and Uncontrolled hypErtension: the DUAL-ICE Pilot Study
Brief Title: Renal Denervation and pUlmonary Vein isolAtion With cryoabLation on Patients With Atrial Fibrillation and hypErtension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUAL-ICE
Record Dates: First submitted 2021-05-17; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-05

CONDITIONS: Paroxysmal Atrial Fibrillation; Hypertension
Keywords: Renal artery cryoablation; Pulmonary vein cryoablation; One-stop cardio-renal combined cryoablation therapy
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Intervention Model Description: Hypertensive patients with symptomatic paroxysmal atrial fibrillation who are to be treated by cryoablation with substandard blood pressure (SBP ≥ 150 mmHg or DBP ≥ 90 mmHg in the clinic with at least one antihypertensive drug)
Who Masked: Participant
Masking Description: We used participant single blindness. To ensure single blindness, femoral artery puncture and renal arteriography were performed in the control group after cryoablation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDN+PVI group (Experimental): The experimental group received renal artery cryoablation and pulmonary vein cryoablation. Pulmonary vein cryoablation was first followed by renal artery cryoablation.
  Interventions: Procedure: Renal artery cryoablation; Procedure: Pulmonary vein cryoablation
- PVI only group (Sham Comparator): The control group received pulmonary vein cryoablation alone. To ensure single blindness, the control group received femoral artery puncture and renal arteriography after cryoablation.
  Interventions: Procedure: Pulmonary vein cryoablation; Procedure: Renal arteriography

INTERVENTIONS:
Procedure: Renal artery cryoablation — Renal denervation were achieved by cryoablation of renal artery with cryoballoon.
  Arms: RDN+PVI group
Procedure: Pulmonary vein cryoablation — Pulmonary vein isolation was achieved by cryoablation of pulmonary veins with cryoballoon.
Procedure: Renal arteriography — Renal artery was examined by renal arteriography
  Arms: PVI only group

SUMMARY:
The DUAL-ICE study is a single-center, prospective, randomized controlled study. The main purpose is to verify that renal artery cryoablation combined with pulmonary vein cryoablation can reduce the recurrence of atrial fibrillation in hypertensive patients with paroxysmal atrial fibrillation and substandard hypertension, and to further verify the clinical significance of one-stop cardio-renal combined cryoablation therapy for hypertension control.

DETAILED DESCRIPTION:
Hypertension is a major risk factor for the high morbidity and mortality of cardiovascular diseases in the world. As a common arrhythmia, the autonomic nervous system plays an important role in the occurrence and maintenance of atrial fibrillation [1,2]. Enhancement of central sympathetic nervous system activity and stimulation of the efferent sympathetic nerve of the heart can promote the occurrence and development of atrial fibrillation [3]. Hypertension is an important risk factor for the occurrence of atrial fibrillation, and the incidence of complications such as heart failure, coronary heart disease and left ventricular hypertrophy is increased in patients with atrial fibrillation with poor blood pressure control [4-6]. Therefore, hypertension management in patients with atrial fibrillation is particularly important.

However, a 2014 study of SYMPLICITY HTN-3 with a sample size of 535 people showed that RDN could not significantly reduce blood pressure [10], which put the study of RDN into a dilemma. Since then, researchers have optimized the study design, and some more detailed results have suggested a significant antihypertensive effect of RDN [11-13].

At present, there are few reports on the cryo-ablation of renal sympathetic nerve in the RDN studies, only the case of cryo-ablation of renal artery by Dr.Prochnau et al in Germany in 2014, which is still a technical blank in China [14]. At present, catheter ablation has been widely recognized in the treatment of paroxysmal atrial fibrillation. In terms of patient comfort and efficacy, cryo-ablation promoted in recent years shows greater advantages than radiofrequency ablation, which has the characteristics of less damage to surrounding tissues and faster recovery of vascular endothelial function. Therefore, the application of cryoablation in the field of RDN may be similar to the effect of pulmonary vein ablation. The purpose of our study was to investigate whether renal artery cryoablation combined with pulmonary vein cryoablation reduces the recurrence rate of atrial fibrillation compared with pulmonary vein cryoablation alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, and <75 years old, gender is not limited;
2. Hypertensive patients with symptomatic paroxysmal atrial fibrillation to be treated by catheter ablation with substandard blood pressure. SBP ≥ 150 mmHg or DBP ≥ 90 mmHg in patients taking at least one antihypertensive drug;
3. Agree to participate and sign the informed consent.

Exclusion Criteria:

1. Cannot accept catheter ablation (such as thrombus in left atrium/left atrial appendage, recent myocardial infarction, stroke, etc.);
2. Patients with obvious bleeding tendency or unable to accept postoperative anticoagulation;
3. The anteroposterior diameter of left atrium indicated by echocardiography was ≥50mm;
4. A history of left atrial surgery or left atrial interventional therapy (including cryo-ablation, radiofrequency ablation, left atrial appendage occlusion, etc.);
5. NYHA grade IV congestive heart failure or LVEF <30%;
6. patients with valvular atrial fibrillation and secondary atrial fibrillation (such as uncontrolled hyperthyroidism, acute alcoholism, atrial fibrillation after cardiac surgery, etc.);
7. Patients with typical atrial fluttering or other supraventricular tachycardia (duration greater than 30s) confirmed by preoperative electrocardiogram or dynamic electrocardiogram;
8. Severe organic heart disease, including moderate to severe mitral insufficiency or stenosis, previous myocardial infarction, hypertrophic cardiomyopathy, etc.;
9. Patients with secondary hypertension;
10. Uncontrollable pulmonary hypertension;
11. Patients with glomerular filtration rate (EGFR) < 45ml/min/1.73m2 or patients with chronic kidney disease, nephrotic syndrome, polycystic kidney disease and other renal diseases were estimated according to MDRD calculation method;
12. Renal artery imaging (renal artery CTA) exclusion criteria:

    1. inability to access the renal vascular system;
    2. Diameter of renal aorta less than 4 mm or length less than 20 mm;
    3. Hemodynamic or anatomical renal artery abnormalities or stenosis;
    4. A history of previous renal artery interventions, including balloon angioplasty or stenting;
    5. There are multiple unilateral renal aortas leading to the kidney;
13. Participated in other clinical studies and not yet enrolled in the group;
14. Women who are pregnant, lactating or preparing to become pregnant;
15. Life expectancy less than 1 year;
16. Other conditions that are not suitable for inclusion in this study as assessed by the researcher, such as mental disorders or psychological disorders;
17. A history of acute coronary events or percutaneous coronary stent intervention, a history of stroke or transient ischemic attack, and extensive atherosclerosis with intravascular thrombosis within the last 6 months;
18. Patients with ICD implantation history or CRT treatment history.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | Within 12 months after procedure (outside the 90-day blanking period).
  Atrial arrhythmia recurrence (documented atrial fibrillation, atrial tachycardia, or atrial flutter for ≥30 seconds during ambulatory monitoring or for ≥10 seconds on a 12-lead ECG), cardioversion, or use of class I or III antiarrhythmic drugs.

SECONDARY OUTCOMES:
Differences in office blood pressure | Within 12 months after procedure.
  Differences in blood pressure (SBP, DBP) between the two groups at 6 and 12 months after procedure compared to the baseline;

OTHER OUTCOMES:
Differences in 24-hour dynamic blood pressure | Within 12 months after procedure.
  The difference of 24h-SBP/DBP mean value (daytime, night and whole day) between the two groups at 6 and 12 months after procedure compared to the baseline level;
Differences in self-measured blood pressure | Within 12 months after procedure.
  Differences in mean self-measured blood pressure (SBP, DBP) from baseline in the two groups at 3, 6, 9 and 12 months after procedure;

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Grassi G. Assessment of sympathetic cardiovascular drive in human hypertension: achievements and perspectives. Hypertension. 2009 Oct;54(4):690-7. doi: 10.1161/HYPERTENSIONAHA.108.119883. Epub 2009 Aug 31. PMID 19720958
- [Background] Schlaich MP, Sobotka PA, Krum H, Whitbourn R, Walton A, Esler MD. Renal denervation as a therapeutic approach for hypertension: novel implications for an old concept. Hypertension. 2009 Dec;54(6):1195-201. doi: 10.1161/HYPERTENSIONAHA.109.138610. Epub 2009 Oct 12. No abstract available. PMID 19822798
- [Background] Arora R, Ng J, Ulphani J, Mylonas I, Subacius H, Shade G, Gordon D, Morris A, He X, Lu Y, Belin R, Goldberger JJ, Kadish AH. Unique autonomic profile of the pulmonary veins and posterior left atrium. J Am Coll Cardiol. 2007 Mar 27;49(12):1340-8. doi: 10.1016/j.jacc.2006.10.075. Epub 2007 Mar 12. PMID 17394967
- [Background] Krahn AD, Manfreda J, Tate RB, Mathewson FA, Cuddy TE. The natural history of atrial fibrillation: incidence, risk factors, and prognosis in the Manitoba Follow-Up Study. Am J Med. 1995 May;98(5):476-84. doi: 10.1016/S0002-9343(99)80348-9. PMID 7733127
- [Background] Benjamin EJ, Levy D, Vaziri SM, D'Agostino RB, Belanger AJ, Wolf PA. Independent risk factors for atrial fibrillation in a population-based cohort. The Framingham Heart Study. JAMA. 1994 Mar 16;271(11):840-4. PMID 8114238
- [Background] Joshi S, Choi AD, Kamath GS, Raiszadeh F, Marrero D, Badheka A, Mittal S, Steinberg JS. Prevalence, predictors, and prognosis of atrial fibrillation early after pulmonary vein isolation: findings from 3 months of continuous automatic ECG loop recordings. J Cardiovasc Electrophysiol. 2009 Oct;20(10):1089-94. doi: 10.1111/j.1540-8167.2009.01506.x. Epub 2009 Jun 22. PMID 19549038
- [Background] Schlaich MP, Sobotka PA, Krum H, Lambert E, Esler MD. Renal sympathetic-nerve ablation for uncontrolled hypertension. N Engl J Med. 2009 Aug 27;361(9):932-4. doi: 10.1056/NEJMc0904179. No abstract available. PMID 19710497
- [Background] Krum H, Schlaich MP, Sobotka PA, Bohm M, Mahfoud F, Rocha-Singh K, Katholi R, Esler MD. Percutaneous renal denervation in patients with treatment-resistant hypertension: final 3-year report of the Symplicity HTN-1 study. Lancet. 2014 Feb 15;383(9917):622-9. doi: 10.1016/S0140-6736(13)62192-3. Epub 2013 Nov 7. PMID 24210779
- [Background] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036
- [Background] Bhatt DL, Kandzari DE, O'Neill WW, D'Agostino R, Flack JM, Katzen BT, Leon MB, Liu M, Mauri L, Negoita M, Cohen SA, Oparil S, Rocha-Singh K, Townsend RR, Bakris GL; SYMPLICITY HTN-3 Investigators. A controlled trial of renal denervation for resistant hypertension. N Engl J Med. 2014 Apr 10;370(15):1393-401. doi: 10.1056/NEJMoa1402670. Epub 2014 Mar 29. PMID 24678939
- [Background] Bohm M, Kario K, Kandzari DE, Mahfoud F, Weber MA, Schmieder RE, Tsioufis K, Pocock S, Konstantinidis D, Choi JW, East C, Lee DP, Ma A, Ewen S, Cohen DL, Wilensky R, Devireddy CM, Lea J, Schmid A, Weil J, Agdirlioglu T, Reedus D, Jefferson BK, Reyes D, D'Souza R, Sharp ASP, Sharif F, Fahy M, DeBruin V, Cohen SA, Brar S, Townsend RR; SPYRAL HTN-OFF MED Pivotal Investigators. Efficacy of catheter-based renal denervation in the absence of antihypertensive medications (SPYRAL HTN-OFF MED Pivotal): a multicentre, randomised, sham-controlled trial. Lancet. 2020 May 2;395(10234):1444-1451. doi: 10.1016/S0140-6736(20)30554-7. Epub 2020 Mar 29. PMID 32234534
- [Background] Kandzari DE, Bohm M, Mahfoud F, Townsend RR, Weber MA, Pocock S, Tsioufis K, Tousoulis D, Choi JW, East C, Brar S, Cohen SA, Fahy M, Pilcher G, Kario K; SPYRAL HTN-ON MED Trial Investigators. Effect of renal denervation on blood pressure in the presence of antihypertensive drugs: 6-month efficacy and safety results from the SPYRAL HTN-ON MED proof-of-concept randomised trial. Lancet. 2018 Jun 9;391(10137):2346-2355. doi: 10.1016/S0140-6736(18)30951-6. Epub 2018 May 23. PMID 29803589
- [Background] Azizi M, Schmieder RE, Mahfoud F, Weber MA, Daemen J, Davies J, Basile J, Kirtane AJ, Wang Y, Lobo MD, Saxena M, Feyz L, Rader F, Lurz P, Sayer J, Sapoval M, Levy T, Sanghvi K, Abraham J, Sharp ASP, Fisher NDL, Bloch MJ, Reeve-Stoffer H, Coleman L, Mullin C, Mauri L; RADIANCE-HTN Investigators. Endovascular ultrasound renal denervation to treat hypertension (RADIANCE-HTN SOLO): a multicentre, international, single-blind, randomised, sham-controlled trial. Lancet. 2018 Jun 9;391(10137):2335-2345. doi: 10.1016/S0140-6736(18)31082-1. Epub 2018 May 23. PMID 29803590
- [Background] Prochnau D, Heymel S, Otto S, Figulla HR, Surber R. Renal denervation with cryoenergy as second-line option is effective in the treatment of resistant hypertension in non-responders to radiofrequency ablation. EuroIntervention. 2014 Sep;10(5):640-5. doi: 10.4244/EIJV10I5A110. PMID 25256203
- [Background] Andrade JG, Wells GA, Deyell MW, Bennett M, Essebag V, Champagne J, Roux JF, Yung D, Skanes A, Khaykin Y, Morillo C, Jolly U, Novak P, Lockwood E, Amit G, Angaran P, Sapp J, Wardell S, Lauck S, Macle L, Verma A; EARLY-AF Investigators. Cryoablation or Drug Therapy for Initial Treatment of Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):305-315. doi: 10.1056/NEJMoa2029980. Epub 2020 Nov 16. PMID 33197159
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Wazni OM, Dandamudi G, Sood N, Hoyt R, Tyler J, Durrani S, Niebauer M, Makati K, Halperin B, Gauri A, Morales G, Shao M, Cerkvenik J, Kaplon RE, Nissen SE; STOP AF First Trial Investigators. Cryoballoon Ablation as Initial Therapy for Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):316-324. doi: 10.1056/NEJMoa2029554. Epub 2020 Nov 16. PMID 33197158
- [Background] Pokushalov E, Romanov A, Corbucci G, Artyomenko S, Baranova V, Turov A, Shirokova N, Karaskov A, Mittal S, Steinberg JS. A randomized comparison of pulmonary vein isolation with versus without concomitant renal artery denervation in patients with refractory symptomatic atrial fibrillation and resistant hypertension. J Am Coll Cardiol. 2012 Sep 25;60(13):1163-70. doi: 10.1016/j.jacc.2012.05.036. Epub 2012 Sep 5. PMID 22958958
- [Background] Steinberg JS, Shabanov V, Ponomarev D, Losik D, Ivanickiy E, Kropotkin E, Polyakov K, Ptaszynski P, Keweloh B, Yao CJ, Pokushalov EA, Romanov AB. Effect of Renal Denervation and Catheter Ablation vs Catheter Ablation Alone on Atrial Fibrillation Recurrence Among Patients With Paroxysmal Atrial Fibrillation and Hypertension: The ERADICATE-AF Randomized Clinical Trial. JAMA. 2020 Jan 21;323(3):248-255. doi: 10.1001/jama.2019.21187. PMID 31961420